CLINICAL TRIAL: NCT05590689
Title: Phase I/II Dose Escalation Trial of Radiodynamic Therapy (RDT) With 5-Aminolevulinic Acid in Patients With First Recurrence of Glioblastoma
Brief Title: Radiodynamic Therapy (RDT) With Gliolan in Patients With First Recurrence of Brain Tumor
Acronym: ALA-RDTinGBM
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: photonamic GmbH & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: WWU20_0041; 2021-004631-92 (EudraCT Number)
Record Dates: First submitted 2022-09-07; First posted 2022-10-21 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Aminolevulinic Acid

STUDY DESIGN:
Intervention Model Description: A modified 3+3 design is used. The maximum tolerated dose of repeated RDT (consisting of 5-ALA dosing an radiotherapy) and safety will be determined in 9 cohorts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiodynamic therapy (RDT) (Experimental): All patients will be treated with RDT. Patients are devided into cohorts which differs in the total amount and frequence of RDT.
  Interventions: Drug: Gliolan; Radiation: Radiodynamic therapy

INTERVENTIONS:
Drug: Gliolan — A repetitive dose of Gliolan will be administrated in combination with radiotherapy (radiodynamic therapy)
  Other Names: 5-Aminolevulinic acid
Radiation: Radiodynamic therapy — Radiotherapy will be performed in combination with Gliolan administration

SUMMARY:
The investigational drug 5-ALA (known under the trade name Gliolan®) is an approved drug for the surgical removal of malignant glioma (WHO grade III and IV). In this trial, the drug is being tested outside of its actual approval as a radiosensitizer in combination with conventional radiotherapy for first-time recurrence (relapse) of malignant glioma. In this clinical trial, the investigational drug 5-ALA is being used for the first time in a multiple dose escalation regimen in combination with radiotherapy following surgical removal of a recurrent malignant glioma in humans. The investigational drug, 5-ALA, has been used as a single dose to date as a standard of care for visualization of malignant tissue in the surgical removal of gliomas.

The planned clinical trial will first and foremost investigate how well repeated administration of the investigational drug 5-ALA is tolerated in combination with radiotherapy. At the same time, the design of the trial serves to optimize this novel therapeutic procedure with regard to the frequency of administration of the investigational drug 5-ALA in combination with radiotherapy for future clinical trials.

As a secondary objective, the efficacy of additional 5-ALA administration will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Written patient consent after comprehensive information
* Age >/= 18 years
* Recurrence of supratentorial glioblastoma after initial resection and adjuvant therapy (e.g. radio-chemotherapy, targeted therapies, antiangiogenic therapies as determined by the tumor board) (with planned second resection cohort 0 and 1), second or third recurrences permitted
* Clinically indicated further radiotherapy as per decision of the tumor board as part of therapy for recurrence
* Histological verification of recurrent glioblastoma independent of methylated MGMT promotor status when alkylating chemotherapy failed at this time.
* Karnofsky Performance Score ≥ 60
* For female and male patients and their female partners of childbearing/reproductive potential(*): Willingness to apply highly effective contraception (Pearl index <1) during the entire study (and for at least 6 months after the first application of 5-ALA). Such methods include:

  1. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation: I. oral II. intravaginal III. transdermal
  2. progestogen only hormonal contraception associated with inhibition of ovulation: I. oral II. injectable III. implantable
  3. intrauterine device (IUD)
  4. intrauterine hormone-releasing system (IUS)
  5. bilateral tubal occlusion
  6. vasectomised partner
  7. male patients have to use a condom
  8. sexual abstinence
* Pre-menopausal(*) female patients with childbearing potential: a negative pregnancy test must be obtained max. 72h prior to treatment start
* Adequate liver function: bilirubin < 1.5 times above upper limit of normal range (ULN), alanine transaminase (ALT/SGPT) and aspartate transaminase (AST/SGOT) < 3 times ULN. In the case of documented or suspected Gilbert's disease bilirubin < 3 times ULN.
* Adequate renal function: creatinine < 3 times above ULN; eGFR >/= 60 ml/min, Blood clotting: INR/Quick/PT and PTT within acceptable limits according to the investigator.

(*) Definition: A man is considered of reproductive potential after puberty unless permanently sterile by bilateral orchidectomy. A woman is considered of childbearing potential (WOCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A post-menopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

* Patient unable to undergo imaging by MRI, PET or contrast-enhanced CT for whatever reason (e.g. pace-maker)
* Pregnant and breastfeeding women
* Past medical history of diseases with poor prognosis, e.g., severe coronary heart disease, heart failure (NYHA III/IV), severe and poorly controlled diabetes, immune deficiency, residual deficits after stroke, severe mental retardation or other serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator)
* Any active infection (at the discretion of the investigator)
* Hypersensitivity against porphyrins
* Known diagnosis of porphyria
* Participation in another clinical trial with therapeutic intervention or use of any other therapeutic interventional agent other than the standard therapy since diagnosis of glioblastoma
* Known intolerance to study medication
* Pre-treatment with other potentially phototoxic or photosensitizing substances (e.g. tetracyclines, sulfonamides, fluoroquinolones, hypericin extracts, products containing St. John's wort ) during the 2 weeks preceding RDT

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 6 weeks after last R(D)T in adjuvant phase
  In the resent study we will investigate the maximum-tolerated dose (MTD) of the combination of 5-ALA and radiation. MTD is defined as the highest number of RDT that does not cause unacceptable side effects, i.e. at which no more than 1 of 6 patients suffers a dose-limiting toxicity (DLT). DLT describes side effects of a drug that are serious enough to prevent an increase of dose (NCI dictionary of cancer terms). In the present study it is defined as any ≥ Gr.3 hematological toxicity, any ≥ Gr.3 neurological toxicity and any ≥ Gr.3 non-hematological toxicity occurring during the 6 week observation period, that does not resolve to pre-treatment baseline or ≤ Gr. 2 within 3 weeks, either spontaneously or with adequate treatment.
  To detect any relevant DLT the following aspects are monitored:
  * Toxicological safety of repeat doses of 5-ALA
  * Neurological safety of RDT
  * Dermatological safety of RDT
  * Assess all new AEs CTCAE grade 2 or higher

SECONDARY OUTCOMES:
Overall survival rate (OSR) | 6 months after first R(D)T in adjuvant phase
  Percentage of patients who are alive 6 months after first R(D)T
progression-free survival rate (PFS) | 6 months after first R(D)T in adjuvant phase
  Percentage of patients without tumor progression 6 months after first R(D)T in adjuvant phase
event-free survival rate (EFS) | 6 months after inclusion
  Percentage of patients without suffering any disease related event such as DLT or progression until 6 months after inclusion
concentration changes of immunhistochemistry marker (e.g. Caspase-3, IBA1, H&E, EvG, P53, Ki 67, gammaH2AX) | during surgery
  analytic results of pharma-radio-dynamic tissue changes. Tissue samples collected during surgery of cohort 0 and 1

OTHER OUTCOMES:
concentration changes of CPI and CPIII | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes as one combined sum parameter
concentration changes of radiobiological marker CD3 | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes
concentration changes of radiobiological marker CD4 | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes
concentration changes of radiobiological marker CD8 | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes
concentration changes of radiobiological marker C19 | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes
concentration changes of radiobiological marker for total leucocyte count | 6 months after first R(D)T in adjuvant phase
  Analytic results for concentration changes

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stummer, Prof. Dr., Principal Investigator — University Hospital Muenster
Locations (1):
- University Hospital Münster, Klinik für Neurochirurgie, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pepper NB, Eich HT, Muther M, Oertel M, Rehn S, Spille DC, Stummer W. ALA-RDT in GBM: protocol of the phase I/II dose escalation trial of radiodynamic therapy with 5-Aminolevulinic acid in patients with recurrent glioblastoma. Radiat Oncol. 2024 Jan 22;19(1):11. doi: 10.1186/s13014-024-02408-7. PMID 38254201